CLINICAL TRIAL: NCT03591198
Title: Improving Health and Reducing Disability of Depressed Elderly With Chronic Conditions Through Qigong Exercise: A Randomized Controlled Trial
Brief Title: Improving Health and Reducing Disability of Depressed Elderly With Chronic Conditions Through Qigong Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor and Head of Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81173316-1
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Chronic Disease; Depressive Symptoms
MeSH Terms: conditions — Chronic Disease; Depression | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Training (Experimental)
  Interventions: Behavioral: Qigong Training
- Cognitive Training (Active Comparator)
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Qigong Training — Eight-Section Brocades
  Arms: Qigong Training
Behavioral: Cognitive Training — Cognitive Training of Memory and Executive Function with Activities requiring Mobilization
  Arms: Cognitive Training

SUMMARY:
Qigong exercise is beneficial for older adults with co-occurring chronic physical illness and depression in terms of psychological and physical outcomes. However, the effects on functional independence, sleep quality, and mobility of depressive older adults remain unclear. It is also important to replicate its benefits for subjective well-being and muscle strength. A randomized clinical trial was conducted among older adults who were aged 60 or above and with chronic medical conditions for one year. After random assignment, intervention group (n = 25) went through qigong exercise twice a week and for 12 weeks,whereas control group (n = 22) was involved in cognitive training activities with mobilization elements. The psychosocial and physical outcomes of the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* have been suffering from chronic medical conditions for more than one year
* have depressive symptoms as indicated by Geriatric Depression Scale (GDS ≥ 6)

Exclusion Criteria:

* have practiced or received training of any form of mind-body exercises (including tai chi, yoga, and qigong) during the 6 months prior to intervention.
* have changed medication or the dosage prior to or during intervention
* have obvious cognitive and language impairment or score less than 20 in Mini-Mental State Examination (MMSE)
* undergo electroconvulsive therapy, psychotherapy, or psychoeducation
* cannot demonstrate satisfactory sitting balance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Personal Well-Being Index (PWI) | the change from baseline to the completion of intervention (12 weeks later)
  It is measured by the 8-item scale of Personal Well-Being Index (PWI). Each item was rated according to an 11-point scale ranging from '0' (extremely dissatisfied) to '10' (extremely satisfied). An overall score of PWI score was the sum of all items. The overall score ranges from 0 to 110, with higher score indicating higher subjective well-being.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured by the 18-item scale of Functional Independence Measure (FIM). Based on a 7-point scale for rating (1 = totally unable; 7 = totally independent), a total score of FIM ranges from 18 to 126 was generated. Higher total score indicates less disability.
Pittsburgh Sleep Quality Index (PSQI) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured by the Pittsburgh Sleep Quality Index (PSQI). It has 19 items measuring 7 components of sleep quality, and a total score is calculated as the sum of all the component scores. The total score ranges from 0 to 21, with lower score showing better sleep quality.
Timed up and Go Test (TUG) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  Timed up and Go Test (TUG) is used to measure mobility. During the test, participants were sitting on a chair, and then they were required to stand up, walk to a mark which is 3 meters away from the chair, go back to the chair from the mark, and sit down again. The time each participant spent to complete the above series of actions was recorded. Participants performed the test for three times, and their final scores were the average of the three. And lower score indicates better mobility.
Handgrip Strength | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured with a Jamar handheld dynamometer. Participants performed three trials of left hand and right hand grip strength, and the final outcome of each hand was calculated as the mean performance of the three trials. Higher score indicates stronger handgrip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechinic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No